CLINICAL TRIAL: NCT03357016
Title: Effect of High-Intensity Interval Training and Moderate-Intensity Continuous Training on Abdominal Fat Mass and Energy Substrates Utilization in Postmenopausal Women
Brief Title: HIIT Versus MICT on Abdominal Fat Mass and Lipid Oxidation in Postmenopausal Women (MATISSE)
Acronym: MATISSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Collaborators: CREPS Vichy Auvergne (Unknown); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AU1303; 2016-A01742-49 (Registry Identifier: ANSM)
Record Dates: First submitted 2017-11-13; First posted 2017-11-29 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2017-12

CONDITIONS: Overweight; Post Menopausal Women
Keywords: interval training; abdominal fat mass; postmenopausal women; lipids oxidation
MeSH Terms: conditions — Overweight | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Masking Description: Data collected on the volunteers will be made anonymous.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training program (HIIT) (Experimental): Subjects perform three sessions of training during 12 weeks: 35 min at 50% maximal aerobic power on bicycle.
  Interventions: Other: Training programs
- Moderate Intensity Continuous Training program (MICT) (Experimental): Subjects perform three sessions of training during 12 weeks: repeated cycles of sprinting for 8s and pedaling slowly for 12s (between 20 and 30 rpm) for a maximum of 60 repeats per session.
  Interventions: Other: Training programs
- HIIT + Resistance Training program (RT) (Experimental): Subjects perform three sessions of training during 12 weeks: Each subject performed HIIT protocol and then a single set of 8 exercises with 1 ou 2min resting period between exercises. Each set consisted of 8-12 repetitions at about 80% maximum repetition.
  Interventions: Other: Training programs

INTERVENTIONS:
Other: Training programs — High Intensity Interval Training program (HIIT) vs. Moderate Intensity Continuous Training program (MICT) vs. High Intensity Interval Training program + Resistance Training program (HIIT+RT)

SUMMARY:
Postmenopausal women, as men, are more prone to central or android obesity than premenopausal women. Abdominal fat mass accumulation is associated with an increase of cardiovascular disease (CVD) risk.

Most exercise programs designed for weight loss have focused on about 30 min several times per week of moderate intensity continuous training (MICT). Disappointingly, such exercise programs have led to either none or low fat loss. Accumulating evidence suggests that high intensity interval training (HIIT) should be an effective exercise protocol for reducing body fat of overweight individuals, especially at the abdominal level.

Resistance Training (RT) is associated with increased muscle mass and strength gain in main muscles groups. Thus, RT seems to be an interesting strategy to fight against deconditioning and autonomy loss with age. Development of muscle mass enhances resting metabolism rate. Thus, RT could raise daily energy expenditure ie. substrates' oxidation including lipids.

The aim of our study was to compare the effects of a 12-week moderate intensity continuous training (MICT) program with high intensity interval training (HIIT) program combined or not with a resistance training (RT) program on total abdominal and visceral fat mass and substrate utilization in postmenopausal women.

It is hypothesized that HIIT compared to MICT program would result in significantly greater whole body and regional fat mass losses (abdominal and visceral) and would improve lipid oxidation at rest and during prolonged moderate exercise. It is also hypothesized that HIIT associated with RT could be the best strategy to reduce fat mass.

DETAILED DESCRIPTION:
Overweight and obesity are dramatically spreading worldwide, and these trends are occurring in both developed and developing countries. Fat mass and more particularly abdominal fat mass is related to the development of cardio-vascular diseases (CVD). Postmenopausal women, as men, are more prone to central or android obesity.

Most exercise programs designed for weight loss have focused on about 30 min several times a week of moderate intensity continuous training (MICT). Disappointingly, such exercise programs have led to either none or low fat losses. Accumulating evidence suggests that high intensity interval training (HIIT) could be an effective exercise protocol for reducing adipose tissue of overweight individuals, especially at the abdominal level. HIIT involves brief high-intensity, anaerobic exercise followed by brief but slightly longer bouts of very low-intensity exercise.

Resistance training (RT) program are currently proposed in order to reduce fat mass / preserve fat-free mass. Their beneficial effects have been demonstrated, especially in the elderly. Through development (or maintenance) of muscle mass, RT increases resting metabolism rate, daily energy expenditure, and substrate (fatty acids) oxidation.

The aim of the study was to compare the effects of a 12-week moderate intensity continuous training (MICT) program with high intensity interval training (HIIT) combined or not with resistance training (RT) program on total, abdominal and visceral fat mass and substrate utilization at rest and during exercise in postmenopausal women.

36 postmenopausal women will be randomly assigned to MICT (n= 12) or HIIT (n= 12) or HIIT + RT (n= 12) group. Subjects performed three sessions per week during 12 weeks, on bicycle.

MICT: For the MICT protocol, each subject performed 35 min at 50% maximal aerobic power (MAP).

HIIT: For the HIIT protocol, each subject performed repeated cycles of sprinting for 8 s and pedaling slowly for 12 s (between 20 and 30 rpm) for a maximum of 60 repeats per session.

HIIT+RT: For the HIIT+RT protocol, each subject performed HIIT protocol. Then they performed a single set of 8 exercises with 1 or 2min resting period between exercises. Each set consisted of 8-12 repetitions at about 80% maximum repetition (MR).

Total body and regional fat content will be measured using dual-energy x-ray absorptiometry (DEXA) before and after the intervention (3 months).

The investigators will examine the effects of HIIT, MICT and HIIT + RT programs on:

* Total fat mass (and appendicular fat mass) (DEXA)
* Total fat free mass (and appendicular fat free mass) (DEXA)
* Glycemic profile (plasma HbA1c, plasma glucose)
* Lipid profile (TG, HDL, LDL, total cholesterol)
* Substrates oxidation at rest and during moderate exercise (40min, 50% of maximal oxygen consumption VO2 max)

Statistical analysis

Appropriate sample size has been calculated given previous results about fat mass loss during HIIT in women and considering the dropouts observed in this type of protocol.

Gaussian distribution of the data will be tested by the Kolmogorov-Smirnov test. Data will be presented as mean ± standard deviation (SD). Comparisons between groups will be made with Mann & Whitney U test or ANOVA when appropriate. Relationships between data will be assessed by Pearson correlation. Significance will be accepted at the p<0.05 level. Statistical procedures will be performed using Statistica software.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (55- 82 years)
* BMI ≥ 25 and < 40
* Able to follow an exercise protocol
* Eating behavior and physical activity stable since at least 3 month

Exclusion Criteria:

* Subject not able to perform exercise after medical examination
* Subject not able to perform bicycle exercise (pains)
* Chronic infection
* Use of β-blocker
* Medical treatment that could interfere with the different outcome measures
* Hormonal Replacement Therapy (HRT)
* Regular consumption of alcohol
* Refusal to sign the consent form

Ages: 55 Years to 82 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline abdominal fat mass (g) after 3 months of training (T3-T0/T0 x 100) | Baseline T0, 3 months after protocol starting
  Total abdominal fat mass will be measured in all patients using DEXA based on the methodology of Martin and Jensen (1991; L1-L2 to pubic rami) before (baseline, T0) and after 3 months of training (T3).

SECONDARY OUTCOMES:
Lipids oxidation evaluated by gas exchange measurements | 1 week, 3 months after protocol starting
  Evolution of lipids oxidation at rest and during prolonged moderate intensity (40min, 50% of VO2max) using an automated gas analysis system. Carbon dioxide (CO2) production and oxygen consumption (CO2) are expressed in L/min. Respiratory exchange ratio is the ratio between CO2 production and O2 consumption (RER = VCO2/VO2).
Visceral fat mass | Baseline T0, 3 months after protocol starting
  Change from baseline in visceral fat mass (g) (estimated from DEXA)
Total fat mass | Baseline T0, 3 months after protocol starting
  Change from baseline in total fat mass (g) (determined from DEXA)
Fat-free mass | Baseline T0, 3 months after protocol starting
  Change from baseline in total fat-free mass (g) (determined from DEXA)
Plasma HbA1c | Baseline T0, 3 months after protocol starting
  Change from baseline in plasma HbA1c
Glucose level | Baseline T0, 3 months after protocol starting
  Change from baseline in plasma glucose measurement
Plasma triglycerides | Baseline T0, 3 months after protocol starting
  Change from baseline in plasma triglycerides
Plasma total cholesterol | Baseline T0, 3 months after protocol starting
  Change from baseline in total cholesterol
Plasma HDL-cholesterol | Baseline T0, 3 months after protocol starting
  Change from baseline in HDL-cholesterol
Plasma LDL-cholesterol | Baseline T0, 3 months after protocol starting
  Change from baseline in LDL-cholesterol
Insulin level | Baseline T0, 3 months after protocol starting
  Change from baseline in plasma insulin measurement

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Pr, Principal Investigator — CHRU Gabriel Montpied Clermont-Ferrand
Locations (1):
- CREPS Vichy Auvergne, Bellerive-sur-Allier, France